CLINICAL TRIAL: NCT02673801
Title: OPtimeret Kirurgisk Visitation af Knæartrose Patienter (OPKVIK)
Brief Title: Optimized Referral of Knee Patients to the Orthopedic Outpatient Clinic
Status: Completed | Type: Observational
Sponsor: Central Jutland Regional Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 63 00001
Record Dates: First submitted 2016-01-22; First posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2015-08

CONDITIONS: Osteoarthritis, Knee
Keywords: Referral and Consultation; Orthopedics
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient referred to orthopedic clinic: Orthopedic assessment in the outpatient clinic as well as a new algorithm (using patient-reported symptoms and radiographic evaluation) will be applied
  Interventions: Other: Orthopedic assessment in the outpatient clinic

INTERVENTIONS:
Other: Orthopedic assessment in the outpatient clinic — Orthopedic assessment based on clinic evaluation, patient symptoms and radiographic evaluation

SUMMARY:
The purpose of the study is to evaluate an algorithm to screen patients with suspected knee osteoarthritis referred to an orthopedic outpatient clinic by using radiographs and patient-reported symptoms. It will be investigated whether the algorithm is able to identify which patients that are deemed relevant to undergo an orthopedic assessment. This will be evaluated by estimating the sensitivity of the new algorithm compared to with the traditional clinical assessment of the patients.

DETAILED DESCRIPTION:
Further description is provided as eligibility criteria and outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a new referral to the orthopedic outpatient clinic with suspected knee osteoarthritis.

Exclusion Criteria:

* Cognitive or language problems that precludes the filling in of the questionnaires
* Unwillingness to answer the questionnaires
* Patients with rheumatoid arthritis, neurological diseases or cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a new referral to the orthopedic outpatient clinic with suspected knee osteoarthritis
Sampling Method: Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
"Relevant" or "Not relevant" for orthopedic assessment | Through study completion, an average of 1 day (at the initial visit in the orthopedic outpatient clinic)
  Results from the algorithm as well as radiographs and the clinic examination

SECONDARY OUTCOMES:
Knee Injury an Osteoarhtritis Outcome Score (KOOS) | At baseline
  Patient reported symptoms, stiffness, pain, activities of daily living (ADL), function in sport and recreation and knee related quality of life

OTHER OUTCOMES:
Kellgren-Lawrence scale | Through study completion, an average of 1 day (at the initial visit in the orthopedic outpatient clinic)
  Radiographic grade of osteoarthritis
Treatment plan | Through study completion, an average of 1 day (at the initial visit in the orthopedic outpatient clinic)
  Evaluated by the orthopedic surgeon
Earlier treatment | At baseline
  Patient-reported

CONTACTS AND LOCATIONS:
Overall Officials: Lone R Mikkelsen, PhD, Principal Investigator — Research physiotherapist
Locations (1):
- Silkeborg Regional Hospital, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: No
Data can be provided upon request, for instance for meta-analysis.